CLINICAL TRIAL: NCT02827097
Title: The Effect of Rectus Sheath Block on the Postoperative Analgesia in the Patients Undergoing Robotic Single Port Cholecystectomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Ji Eun Kim, Assistant professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AJIRB-MED-CT4-16-127
Record Dates: First submitted 2016-07-04; First posted 2016-07-11 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Gallbladder Diseases
MeSH Terms: conditions — Gallbladder Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Rectus sheath block group (Experimental): 1. administration of denogan
  2. rectus sheath block with 0.375% ropivacaine
  Interventions: Drug: denogan and rectus sheath block
- Control group (Placebo Comparator): just administration of denogan
  Interventions: Drug: denogan

INTERVENTIONS:
Drug: denogan and rectus sheath block — administration of denogan and rectus sheath block with 0.375% ropivacaine
  Arms: Rectus sheath block group
Drug: denogan — administration of denogan
  Arms: Control group

SUMMARY:
The primary purpose of this study is to investigate the effect of rectus sheath block on abdominal pain score after robotic single port cholecystectomy.

The secondary purpose of this study is to investigate the effect of rectus sheath block on fentanyl consumption during stay of recovery room after surgery.

ELIGIBILITY:
Inclusion Criteria:

* robotic single Port cholecystectomy for gallbladder disease

Exclusion Criteria:

* Allergy to ropivacaine, infection, history of abdominal surgery, body mass index more than 30

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Abdominal pain score after surgery | Change from baseline abdominal pain score up to 24 hours

SECONDARY OUTCOMES:
Fentanyl consumption in recovery room | Up to 1 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Ajou University School of Medicine, Suwon, Seoum, South Korea